CLINICAL TRIAL: NCT06407232
Title: An Interventional Study of Letermovir for Secondary Prophylaxis After Treatment of Cytomegalovirus Infection in High Risk (D+/R-) Kidney and Kidney/Pancreas Transplant Recipients
Brief Title: Letermovir (Prevymis) for CMV in Kidney and Pancreas Transplant Recipients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0174; A561000 (Other: UW Madison); Protocol Version 8/22/25 (Other: UW Madison); 235208 (Other: OnCore ID)
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Cytomegalovirus Infections; Kidney Transplant Infection; Pancreas Transplant
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — letermovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Letermovir for CMV in Transplant Patients (Experimental): Enrolled participants will be converted from treatment with ganciclovir derivatives to letermovir
  Interventions: Drug: Letermovir

INTERVENTIONS:
Drug: Letermovir — 480 mg taken orally once daily, for 84 days
  Other Names: Prevymis

SUMMARY:
This study is designed to assess how effective letermovir is in preventing recurrence of cytomegalovirus (CMV) infection in adult kidney or kidney/pancreas transplant recipients who are UW Health patients. Participants will be in the study for about 6 months.

DETAILED DESCRIPTION:
Study Population: Patients over 18 years of age who have undergone kidney or simultaneous kidney/pancreas transplant and are high-risk CMV serostatus (D+/R-) at time of transplant who develop CMV viremia that necessitates treatment per our institutional protocol (enrolled in our CMV stewardship monitoring initiative) and demonstrate proven or presumptive lack of cell-mediated immunity, either by CMI testing or risk factor screening.

Patients will be converted from treatment with ganciclovir derivatives to letermovir (480 mg tablet taken orally once daily) when the viral load via standard of care (SOC) weekly monitoring is < 500 IU/mL. This differs from SOC which only allows conversion to secondary prophylactic treatment after CMV is no longer detected on polymerase chain reaction (PCR) for 2 consecutive weeks. Thus, liberalization of conversion threshold will allow for reduced exposure to valganciclovir via reduced duration of therapy allowing relief of the myelosuppressive toxicity and creates an environment conducive to cell-mediated immunity (CMI).

The primary objective is to assess the efficacy of letermovir as secondary prophylaxis after treatment of CMV infection.

The secondary objective is to detect the development of cytomegalovirus-specific cell-mediated immunity as determined by a positive result using the Eurofins-Viracor CMV inSIGHTTM T Cell Immunity Testing per manufacturer specifications.

ELIGIBILITY:
Inclusion Criteria:

* undergone kidney or simultaneous kidney/pancreas transplant
* high-risk CMV serostatus (D+/R-) at time of transplant
* develop CMV viremia that necessitates treatment per our institutional protocol (enrolled in the CMV stewardship monitoring initiative)
* demonstrate proven or presumptive lack of CMI, either by CMI testing or risk factor screening
* able to provide informed consent to participate

Exclusion Criteria:

* contraindication to letermovir or its excipients
* develop ganciclovir-resistant CMV infection
* currently participating in any study involving the administration of a CMV vaccine or another CMV investigational agent
* unable or unwilling, in the opinion of the Investigator, to comply with the protocol
* pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of distinct episodes of any cytomegalovirus replication greater than 1000 IU/mL | up to 90 days after withdrawal of secondary prophylaxis (up to 6 months on study)
  To test the hypothesis that letermovir will be associated with reduced incidence of recurrent viremia, recurrence will be measured defined as incidence of any cytomegalovirus replication greater than 1000 IU/mL requiring treatment after withdrawal of secondary prophylaxis.
Duration of valganciclovir (VGC) Treatment | up to 2 months
  To test the hypothesis that letermovir will be associated with reduced duration of (val)ganciclovir treatment, the duration of VGC treatment will be measured.

SECONDARY OUTCOMES:
Number of Participants with Positive Result for T-Cell Immunity Panel (TCIP) Testing | letermovir initiation (Day 0), at secondary prophylaxis completion (Week 12 +/- 28 days)
  To test the hypothesis that letermovir will be associated with increased development of cytomegalovirus-specific cell-mediated immunity when compared to a literature-based control, development of cytomegalovirus-specific cell-mediated immunity as determined by a positive result using the Eurofins-Viracor CMV inSIGHTTM T-Cell Immunity Testing per manufacturer specifications will be measured.
  TCIP will be collected from the medical record at these timepoints if possible. Given SOC, access to this test is not always available to all patients at both timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Sandesh Parajuli, MBBS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No